CLINICAL TRIAL: NCT02609997
Title: Comparison of In-the-bag Stability Between Single-piece and Three-piece Intraocular Lens Via Scheimpflug Imaging System
Brief Title: Comparison of In-the-bag Stability Between Single-piece and Three-piece Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Home for Cataract Children, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCPMOH2010-China9
Record Dates: First submitted 2015-11-14; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Cataract
Keywords: Intraocular lens
MeSH Terms: conditions — Cataract | interventions — Drug Implants; proxymetacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-piece IOL Group (Experimental): Age-related cataract patients receive in-the-bag implantation of a single-piece IOL
  Interventions: Procedure: Phacomulsification lens removal cataract surgery with single-piece Intraocular lens(IOL) implantation; Drug: Subconjunctival dexamethasone; Device: Viscoelastic materials; Drug: proparacaine
- Three-piece IOL Group (Experimental): Age-related cataract patients receive in-the-bag implantation of a three-piece IOL
  Interventions: Procedure: Phacomulsification lens removal cataract surgery with three-piece Intraocular lens(IOL) implantation; Drug: Subconjunctival dexamethasone; Device: Viscoelastic materials; Drug: proparacaine

INTERVENTIONS:
Procedure: Phacomulsification lens removal cataract surgery with single-piece Intraocular lens(IOL) implantation — The phacoemulsification lens removal cataract surgery is performed with single-piece IOL.During Phacoemulsification.
  Arms: Single-piece IOL Group
Procedure: Phacomulsification lens removal cataract surgery with three-piece Intraocular lens(IOL) implantation — The phacoemulsification lens removal cataract surgery is performed with three-piece IOL.During Phacoemulsification.
  Arms: Three-piece IOL Group
Drug: Subconjunctival dexamethasone — All patients received subconjunctival dexamethasone (2 mg) during surgery. Topical anesthesia, consisting of a single drop of 0.5% proparacaine (Alcaine, Alcon Laboratories), was administered three times at intervals of 5 minutes prior to surgery
Device: Viscoelastic materials — viscoelastic materials are used to protect corneal endothelial cells
Drug: proparacaine — 0.5% proparacaine (Alcaine, Alcon Laboratories)

SUMMARY:
Rapid advances of cataract surgery techniques and intraocular lens (IOL) technology have enabled the transition of cataract surgery from blindness relief to refractive correction. An ideal IOL is the critical component to achieve the refractive target of cataract surgery. Biocompatibility, rate of posterior capsule opacification (PCO) and visual quality have all been suggested as the critical factors of an ideal IOL and widely investigated. Recently, stability of IOL position has also been suggested as one of those critical factors due to its close correlation with postoperative visual function. Data suggests that IOL forward movement of 0.29 mm along the visual axis is associated with -0.4D myopic shift. Wang and colleagues recently reported that 0.5mm decentration of an aspheric IOL could eliminate its aberration-correcting effect. Poor stability could even lead to IOL exchange, an additional surgery that put both surgeons and patients in pain.

As the supporting element of an IOL, the haptics are crucial to keep the IOL in place. Various haptic designs are being compared in terms of position stability of IOLs. Haptic designs of single-piece versus 3-piece are often compared because they are currently the most commonly used types. Single-piece IOLs have soft and broader haptics which are made of the same material as the optic, usually hydrophobic or hydrophilic acrylic, whereas 3-piece IOLs have rigid haptics which are made of poly methyl methacrylate (PMMA). Clinical studies comparing these haptic designs have yielded controversial results regarding their position stability in the capsular bag, which is the most recommended site for IOL fixation in an uneventful cataract surgery.

DETAILED DESCRIPTION:
Rapid advances of cataract surgery techniques and intraocular lens (IOL) technology have enabled the transition of cataract surgery from blindness relief to refractive correction. An ideal IOL is the critical component to achieve the refractive target of cataract surgery. Biocompatibility, rate of posterior capsule opacification (PCO) and visual quality have all been suggested as the critical factors of an ideal IOL and widely investigated. Recently, stability of IOL position has also been suggested as one of those critical factors due to its close correlation with postoperative visual function. Data suggests that IOL forward movement of 0.29 mm along the visual axis is associated with -0.4D myopic shift. Wang and colleagues recently reported that 0.5mm decentration of an aspheric IOL could eliminate its aberration-correcting effect. Poor stability could even lead to IOL exchange, an additional surgery that put both surgeons and patients in pain.

As the supporting element of an IOL, the haptics are crucial to keep the IOL in place. Various haptic designs are being compared in terms of position stability of IOLs. Haptic designs of single-piece versus 3-piece are often compared because they are currently the most commonly used types. Single-piece IOLs have soft and broader haptics which are made of the same material as the optic, usually hydrophobic or hydrophilic acrylic, whereas 3-piece IOLs have rigid haptics which are made of poly methyl methacrylate (PMMA). Clinical studies comparing these haptic designs have yielded controversial results regarding their position stability in the capsular bag, which is the most recommended site for IOL fixation in an uneventful cataract surgery.

Most previous studies measure the IOL position based on Purkinje reflections. The measurement is time-consuming and patients are reluctant to cooperate during image acquisition. Purkinje measurement does not detect anterior chamber depth (ACD) and as such cannot reveal the IOL position along the axis. Clinical Scheimpflug systems based on rotating Scheimpflug imaging, on the other hand, is able to acquire sufficient 3-dimensioinal data points within a reasonably short period, usually seconds. It was shown that these systems are one of the best methods to estimate IOL position. To better compare the intracapsular stability between single-piece and 3-piece IOLs, the investigators measured IOL positions with rotating Scheimpflug imaging systems and tested the visual quality of patients implanted with these IOLs.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bilateral age-related cataract and age between 60 to 85 years

Exclusion Criteria:

* vision-impairing diseases other than cataract, severe refractive error (Preoperative spherical equivalent of either eye >-6.00D or +5.00D)
* history of ocular trauma, past refractive surgery or other ophthalmic surgery, capsular or zonular disorders that might affect the post-operative centration of IOLs
* surgical complications including severe hyphema, iris injury, repeated IOL implantation
* unable to achieve in-the-bag implantation of IOL, corneal sutures during surgery

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The grade of in-the-bag stability between single-piece intraocular lenses (IOLs) and three-piece intraocular lenses(IOLs) | 3 months after the surgery

SECONDARY OUTCOMES:
The visual acuity between single-piece intraocular lenses (IOLs) and three-piece intraocular lenses(IOLs) | 3 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Korynta J, Bok J, Cendelin J. Changes in refraction induced by change in intraocular lens position. J Refract Corneal Surg. 1994 Sep-Oct;10(5):556-64. PMID 7530106
- [Background] Wang L, Koch DD. Effect of decentration of wavefront-corrected intraocular lenses on the higher-order aberrations of the eye. Arch Ophthalmol. 2005 Sep;123(9):1226-30. doi: 10.1001/archopht.123.9.1226. PMID 16157803
- [Background] Rosales P, Marcos S. Phakometry and lens tilt and decentration using a custom-developed Purkinje imaging apparatus: validation and measurements. J Opt Soc Am A Opt Image Sci Vis. 2006 Mar;23(3):509-20. doi: 10.1364/josaa.23.000509. PMID 16539046
- [Background] de Castro A, Rosales P, Marcos S. Tilt and decentration of intraocular lenses in vivo from Purkinje and Scheimpflug imaging. Validation study. J Cataract Refract Surg. 2007 Mar;33(3):418-29. doi: 10.1016/j.jcrs.2006.10.054. PMID 17321392
- [Derived] Zhong X, Long E, Chen W, Xiang W, Liu Z, Chen H, Chen J, Lin Z, Lin H, Chen W. Comparisons of the in-the-bag stabilities of single-piece and three-piece intraocular lenses for age-related cataract patients: a randomized controlled trial. BMC Ophthalmol. 2016 Jul 8;16:100. doi: 10.1186/s12886-016-0283-4. PMID 27392024
- See also: Description Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/